CLINICAL TRIAL: NCT02755857
Title: A Single-arm, Multiple-Dose, Steady-State, Bioavailability Study With Twice Daily Dosing of Lozanoc™ (65 mg Itraconazole Capsules, Mayne) Taken Regardless of Food
Brief Title: Bioavailability Study of Lozanoc™ 65 mg Itraconazole Capsules in Patients Requiring Prophylaxis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayne Pharma International Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MPG011
Record Dates: First submitted 2016-04-28; First posted 2016-04-29 (Estimated); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Neutropenia
Keywords: Prophylaxis; Bioavailability; Pharmacokinetics
MeSH Terms: conditions — Neutropenia | interventions — Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lozanoc (Experimental): 65 mg, capsules, at least 2 capsules twice a day
  Interventions: Drug: Lozanoc

INTERVENTIONS:
Drug: Lozanoc — 65 mg
  Other Names: itraconazole

SUMMARY:
This open-labelled, single arm study is a follow-on from Study MPG010 to compare the relative bioavailability of Lozanoc 65 mg Capsules against Lozanoc 50 mg Capsules and Sporanox 100 mg Capsules in patients requiring itraconazole anti-fungal prophylaxis.

DETAILED DESCRIPTION:
After confirmation of eligibility, participants will take their last dose of current itraconazole therapy (Lozanoc 50mg capsules or Sporanox 100mg capsules) on the morning of Day 1, and commence therapy with Lozanoc 65 mg capsules for 21 days from the evening of Day 1.

The number of Lozanoc 65mg capsules to be taken by the participant will be 2 capsules (130mg) morning and evening OR the same number of Lozanoc 50mg capsules that the participant received in study MPG010, if applicable. That is, if the participant received 3 x 50mg Lozanoc capsules morning and evening on study MPG010 he/she will receive 3 x 65 mg Lozanoc 65 mg capsules, morning and evening in study MPG011

The dose of study drug (Lozanoc 65mg) may be dose-reduced or ceased for toxicity at the discretion of the investigator.

Participants will undergo the following assessments during the course of the study:

* Concurrent medication(s)
* Clinical adverse events
* Measurement of vital signs (weight, blood pressure, temperature)
* Targeted physical examination
* Documentation of any evidence of systemic fungal infection
* Medication and meal diaries
* 12-lead electrocardiogram (ECG)
* Laboratory safety assessments

  * Renal function and electrolytes (urea, creatinine, estimated glomerular filtration rate [eGFR], sodium, potassium, chlorine, bicarbonate)
  * Liver function tests (bilirubin, albumin, total protein, alanine aminotransferase [ALT], aspartate aminotransferase [AST])
* Pharmacokinetic testing

  * pre-morning dose (0 h sample) at Baseline (Day 1), and at Days 8, 15, and 22
  * at 2, 3.5 and 6 hours post the morning dose at Baseline (Day 1) and Day 22

ELIGIBILITY:
Inclusion Criteria:

* Provision of written, informed consent
* Age of at least 18 years
* No clinical evidence of active systemic fungal infection
* Physician-recommended continuation of oral itraconazole as primary prophylaxis in patients at risk of systemic fungal infections or otherwise requiring a long-term itraconazole maintenance regimen, including patients:

  * who have had or are about to have a heart, lung or bone marrow transplant
  * on combination chemotherapy for cancer
  * with an aspergilloma, chronic pulmonary aspergillus bronchitis, or allergic bronchopulmonary aspergillosis
* At least 21 days of prior dosing with oral itraconazole, either Lozanoc 50mg capsules twice daily or Sporanox 100mg capsules twice daily.
* Body mass index between 15.0 and 35.0 kg/m2

Exclusion Criteria:

* Pregnant, planning pregnancy or breastfeeding
* Plasma itraconazole concentration greater than 1500ng/mL (in patients on Lozanoc 50mg capsules)
* Congestive cardiac failure or other causes of ventricular dysfunction that may outweigh the benefit of itraconazole
* Hypersensitivity to Lozanoc or to any of its excipients
* Coadministration of the following drugs:

  * CYP3A4 metabolised substrates that can prolong the QT-interval: sertindole, terfenadine
  * CYP3A4 metabolised 3-hydroxy-3-methylglutaryl-coenzyme A (HMG-CoA) reductase inhibitors: simvastatin, lovastatin
  * Potent CYP3A4 inhibitor: dronedarone
  * Triazolam, alprazolam and oral midazolam
  * Ergot alkaloids such as dihydroergotamine, ergometrine (ergonovine) and ergotamine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Steady-state plasma itraconazole concentrations | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Marriott, MBBS BSc(MED) FRACP FRCPA, Principal Investigator — St Vincent's Hospital
Locations (1):
- St Vincent's Hospital, Darlinghurst, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No
Individual patient data will not be made available